CLINICAL TRIAL: NCT01348282
Title: Exploratory Controlled Prospective Randomized Trial to Compare the Efficacy and Safety of Two Different Pharmacology Strategies on Neurocognitive Impairment in HIV Infection. The TRIANT-TE Study
Brief Title: Efficacy and Safety of Two Pharmacologic Strategies on Neurocognitive Impairment in HIV Infection. The TRIANT-TE Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIANT-TE
Record Dates: First submitted 2011-04-18; First posted 2011-05-05 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Neurocognitive Disturbance; HIV Infection
Keywords: Neurocognitive Impairment; Controlled Randomized Trial; Coadjunctive Treatments; Lithium; Rivastigmine; Antiretroviral Therapy; HIV Infection
MeSH Terms: conditions — Cognition Disorders; HIV Infections | interventions — Lithium; Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lithium (Experimental): Lithium group: Patients who will initiate therapy with lithium, in tablets, beginning a 2-daily 400 mg dose, and changing further adjusting the dose according to drug levels in serum.
  Interventions: Drug: Lithium
- Rivastigmine (Active Comparator): rivastigmine, in transdermal patch administration, beginning a once-daily 4.6 mg dose, and changing further increasing the dose up to once-daily 9.5 mg.
  Interventions: Drug: Rivastigmine
- Control group (No Intervention): Patients who will not initiate treatment

INTERVENTIONS:
Drug: Lithium — lithium, in tablets, beginning a 2-daily 400 mg dose, and changing further adjusting the dose according to drug levels in serum.
  Arms: Lithium
Drug: Rivastigmine — rivastigmine, in transdermal patch administration, beginning a once-daily 4.6 mg dose, and changing further increasing the dose up to once-daily 9.5 mg.
  Arms: Rivastigmine

SUMMARY:
The current project proposes the comparison of two pharmacologic strategies as adjunctive treatments for the improvement of HIV-associated neurocognitive disruption, additionally to use of HAART. The investigators propose the use of the compound that has shown greatest benefits in this context to date, the lithium, versus the use of a well-tolerated and promising drug in other pathologies with neurocognitive affectation, such as Alzheimer or Parkinson diseases, which is the rivastigmine. In those other diseases, this second compound has recently offered a good tolerability, but also benefits on attention, memory and other neurocognitive areas. Both study groups, patients on therapy with lithium and patients on therapy with rivastigmine, will be compared to a control group, which will not initiate any other treatment (therefore only continuing antiretroviral therapy). The investigators are aware that this proposal will offer new relevant data for the study of neurocognitive improvement in HIV infection, as well will allow a better knowledge of clinical management of HIV-infected patients with CNS disease, an aspect that is a common clinical concern today.

DETAILED DESCRIPTION:
Adjunctive treatments based on neurocognitive improvement for HIV-infected patients with CNS disruption have consisted essentially of neurostimulant or neuroprotective treatments. Reports published to date have involved valproic acid, peptide T, CPI-1189, selegiline, memantine, minocycline and lithium. Regarding valproic acid, two trials have confirmed lack of benefit using this compound on HIV-associated neurocognitive decline. In case of peptide T, CPI-1189, selegiline, memantine and minocycline, although their potential mechanisms on brain follow different pathways, trend towards improvement on neurocognitive functioning has been observed. Nonetheless, results on those trials are particularly based on a short term and, moreover, mild connections with benefits on neurocognitive and functional measures have been established. The lithium has been the compound showing clearest benefits on this regard. Two reports have consistently demonstrated benefits on neurocognitive performance using this neuroprotective agent, both in patients with HIV and showing impairment previously. However, lithium is well known to be a drug not easily incorporated in routine practice, at least further than in a psychiatry context. In addition, adverse events related to their use are relatively frequent, and therefore clinical follow-up must be especially controlled. Besides, lithium concentrations are also a concerning aspect considering its use, and drug plasma levels are recommended to be performed throughout the therapy application.

For all these reasons, the current project proposes the comparison of two pharmacologic strategies as adjunctive treatments for the improvement of HIV-associated neurocognitive disruption, additionally to use of HAART. The investigators propose the use of the compound that has shown greatest benefits in this context to date, the lithium, versus the use of a well-tolerated and promising drug in other pathologies with neurocognitive affectation, such as Alzheimer or Parkinson diseases, which is the rivastigmine. In those other diseases, this second compound has recently offered a good tolerability, but also benefits on attention, memory and other neurocognitive areas. Furthermore, in the case of this project, rivastigmine is suggested to be used through a transdermal system patch, a fact that can provide suitability and comfortability with regard to the selected administration method. Both study groups, patients on therapy with lithium and patients on therapy with rivastigmine, will be compared to a control group, which will not initiate any other treatment (therefore only continuing antiretroviral therapy). The investigators are aware that this proposal will offer new relevant data for the study of neurocognitive improvement in HIV infection, as well will allow a better knowledge of clinical management of HIV-infected patients with CNS disease, an aspect that is a common clinical concern today.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 20 to 75 years old
* Correct understanding of study objectives
* Written consent signed
* HIV infection confirmed by Western Blot or two ELISA tests
* Existence of an HIV-associated neurocognitive disorder according to the diagnosis classification offered by Antinori and cols (Neurology, 2007)
* Being on antiretroviral treatment.
* Spanish/Catalan speaker.

Exclusion Criteria:

* To be on a treatment that may interact pharmacologically with any of the new drugs used in study arms.
* Breastfeeding, pregnancy or fertile women willing to be pregnant.
* Renal failure or severe cardiovascular disease.
* Weakness, dehydration or severe sodium depletion.
* Sick sinus syndrome or cardiac conduction disturbances (sinoatrial block or atrioventricular block).
* Active duodenal or gastric ulcer.
* Urinary obstruction.
* Epilepsy.
* Chronic obstructive pulmonary disease (COPD).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Percentage of persons with neurocognitive impairment in the different study groups | From screening to month 12
  The main variable to consider is the existence of HIV-associated neurocognitive impairment. Therefore, the percentage of persons with neurocognitive impairment in different study groups will be the main variable that will report on the improvement associated with new treatments.

SECONDARY OUTCOMES:
Adverse events associated with the initiation of therapy and toxicity parameters | Week 2, month 1, 3, 6, 9, 12
Emotional variables | Baseline, month 3, 6, 12.
  Depression and anxiety symptoms will be assessed by HADS questionnaire.
Functional variables | Baseline, month 3, 6, 12.
  A total of six scales assessing functional interference regarding activities of daily living, as well as self-reported neurocognitive functioning, will be measured.
Quality of life variables | Baseline, month 3, 6, 12.
  Four dimensions concerning quality of life, evaluated by MOS-HIV questionnaire, and satisfaction scales, based on treatments and clinical status, will be evaluated.
Demographics | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació LLuita contra la SIDA, Badalona, Barcelona, Spain